CLINICAL TRIAL: NCT02477761
Title: Sustained Effects of a Non-glucidic Nutrient Preload on Glucose Tolerance in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Andrea Natali, Prof., Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LisbLungo
Record Dates: First submitted 2015-06-17; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water preload (No Intervention): During the "Water preload" study, each subject consume 500 ml of water 30 minutes before a 75 g glucose ingestion
- Nutrient preload (Experimental): During the "Nutrient preload" study, each subject consume a small mixed meal 30 minutes before a 75 g glucose ingestion. The meal is composed by 50 g of parmesan cheese, one small size boiled egg and 300 ml of water (250 kcal, 23 g protein, 17 g fat and 2 g of carbohydrate).
  Interventions: Dietary Supplement: Nutrient preload

INTERVENTIONS:
Dietary Supplement: Nutrient preload — Ingestion of a small mixed protein and lipid meal 30 minutes before glucose
  Arms: Nutrient preload

SUMMARY:
The investigators aimed at evaluating the effects of a small non-glucidic nutrient preload on plasma glucose, insulin, C-peptide, glucagon-like peptide-1, and glucose-dependent insulinotropic polypeptide concentrations after the meal consumption and for 300 min after a 75 g glucose ingestion in diet-controlled type 2 diabetic patients.

DETAILED DESCRIPTION:
As supported by experimental and clinical data, oral carbohydrate tolerance is influenced by the coingestion of nutrients through multiple mechanisms. The ingestion itself, the contact with the gastric mucosa, the arrival into the intestine and the subsequent digestion are known to produce neural reflexes, hormonal responses and plasma substrates gradients which, by modulating gastric emptying, insulin secretion and insulin clearance participate in the regulation of postprandial glycaemia. The size of this effect is influenced by a number of factors: the specific nutrient chemical characteristics (fat vs protein and composition) and their physical properties (solid vs liquid), the timing (pre-load vs coingestion) and finally the individual glucose tolerance status. The effect on 5 h glucose excursions of a combination of protein and fat given before carbohydrate is still unknown.

ELIGIBILITY:
Inclusion Criteria:

* Diet-controlled type 2 diabetic patients
* Subjects ≥ 18 and ≤65 years of age
* Lean, Overweight or Obese (BMI: 18 to 35 kg/m2)
* Normal liver and kidney function
* Normal thyroid function
* Read and understood the informed consent form and signed it voluntarily

Exclusion Criteria:

* Liver, heart, kidney, lung, infectious, neurological, psychiatric, immunological or neoplastic diseases.
* Type 1 or insulin treated diabetes.
* Pregnancy or lactation
* Illicit drug abuse or alcoholism
* Subjects taking anoretic drugs
* Subjects on steroid treatment
* Subjects after bariatric surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose concentration | 330 minutes

SECONDARY OUTCOMES:
Plasma Insulin concentration | 330 minutes
Plasma C-peptide concentration | 330 minutes
Plasma glucagon-like peptide-1 concentration | 330 minutes
Plasma glucose-dependent insulinotropic polypeptide concentration | 330 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natali, Prof, Study Chair — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy